CLINICAL TRIAL: NCT04459598
Title: An Open-label, Parallel Drug Interaction Study to Evaluate the Effect of a CYP3A Moderate Inducer Efavirenz on the Pharmacokinetics of Quizartinib in Healthy Subjects
Brief Title: A Study of the Effect of a Moderate CYP3A Inducer Efavirenz on Quizartinib Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC220-A-U106
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Healthy Subjects; Drug-drug Interaction; Pharmacokinetics; Quizartinib
Keywords: Healthy Subjects; Drug-drug Interaction; Pharmacokinetics; Quizartinib; CYP3A Inducer
MeSH Terms: interventions — efavirenz; quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efavirenz 600 mg + Quizartinib 60 mg (Experimental): Participants who received efavirenz 600 mg once daily (QD) for 34 days and a single, oral dose of quizartinib 60 mg on Day 15 concurrently with efavirenz.
  Interventions: Drug: Efavirenz; Drug: Quizartinib
- Quizartinib 60 mg (Active Comparator): Participants who received a single, oral dose of quizartinib 60 mg on Day 1.
  Interventions: Drug: Quizartinib

INTERVENTIONS:
Drug: Efavirenz — Single oral dose, 600-mg tablet
  Arms: Efavirenz 600 mg + Quizartinib 60 mg
Drug: Quizartinib — Single oral dose, 60 mg (2 x 30 mg) tablets

SUMMARY:
This drug-drug interaction (DDI) study has been designed to investigate the effect of a moderate CYP3A inducer efavirenz on the pharmacokinetics of quizartinib and its major circulating active metabolite AC886.

DETAILED DESCRIPTION:
In vitro, quizartinib is metabolized primarily by CYP3A. Therefore, co-administration of quizartinib with CYP3A inducers may decrease quizartinib exposure. This study will assess the effect of a moderate CYP3A inducer efavirenz on the single dose (60 mg) quizartinib pharmacokinetics in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 to 55 years of age (inclusive), with a body mass index (BMI) of 18 kg/m^2 to 32 kg/m^2 (inclusive) and with a minimum body weight of 45 kg at Screening.
* In females, documented surgical sterilization, postmenopausal status for at least 1 year (follicle stimulating hormone [FSH] > 40 mIU/mL serum at Screening), or agreement to use an approved form of contraception
* In males, agreement to avoid sperm donation for 6 months days after the dose of quizartinib
* Participants must agree to refrain from donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, and platelets from 6 weeks prior to Screening.
* Liver function test results must be below the upper limit of normal. Hemoglobin levels must be ≥ 11.5 g/dL for female participants and ≥ 12.5 g/dL for male participants.
* All participants must be willing to refrain from consuming grapefruit/ grapefruit juice, Seville oranges, and pomegranates/pomegranate juice 10 days before the dose of the study drug is given on Day 1 until end-of-study.

Exclusion Criteria:

* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormality) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Laboratory results (serum chemistry, hematology, and urinalysis) outside the normal range, if considered clinically significant by the investigator. Estimated glomerular filtration rate (eGFR) < 90 mL/min at screening.
* Women who are pregnant or breastfeeding
* Use of any drugs or substances known to be inhibitors or inducers of CYP3A4/5 within 28 days from the first dose or 5 half-lives, if known, of the drugs or substances, whichever is greater, prior to quizartinib administration and during the study.
* Receipt of any prescribed or over-the-counter (OTC) systemic, herbal (including St John's wort), or topical medication within 14 days of quizartinib administration, or any expectation of requiring use of such medication while participating in the study is prohibited.
* Presence or history of clinically severe adverse reaction to any drug
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (with the exception of appendectomy, hernia repair, and/or cholecystectomy)
* History of any cancer, except non-melanoma skin cancer, or resected nonmetastatic cancer with no evidence of disease accepted by the Investigator and Sponsor medical monitor
* A positive drugs of abuse screen from a urine ethanol test (unless the drug is medically prescribed by a licensed health care provider) or alcohol breath test at Screening or at Check-in on Day -1 or a participant who will not agree to smoke ≤10 cigarettes or equivalent per day from Screening up to Enrollment, and is unable to be restricted to ≤5 cigarettes per day and for 6 hours post dose during their period of residence in the clinical unit
* Concomitant use of medications known to affect the elimination of serum creatinine (e.g., trimethoprim or cimetidine) and inhibitors of renal tubular secretion (eg, probenecid) within 14 days or 5 half-lives, if known, of the drugs, whichever is greater, prior to quizartinib administration
* History or presence of an abnormal electrocardiogram (ECG), which, in the investigator's opinion, is clinically significant and/or a QT interval corrected for heart rate using Fridericia's formula >450 milliseconds (ms) at Screening.
* Use of drugs with a risk of QT interval prolongation or torsade de pointes within 14 days of Day -1 (or 5 drug half-lives, if 5 drug half-lives are expected to exceed 14 days)
* Consumption of alcohol- and caffeine-containing beverages within 72 h prior to check-in and during confinement
* Positive serology for hepatitis B surface antigen (HBsAg) and HCV (healthy participants), hepatitis A virus (HAV) immunoglobulin M, or antihuman immunodeficiency virus (HIV) Type 1 and Type 2 (all subjects)
* Loss of more than 450 mL blood during the 3 months before the trial (eg, as a blood donor)
* Current enrollment in or have not yet completed at least 30 days or 5 elimination half-lives, whichever is longer, since receiving an investigational device or product, or receipt of other investigational agents within 30 days of quizartinib

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 participants who met all inclusion criteria and no exclusion criteria were enrolled from 19 Aug 2020 to 14 Oct 2020 at 1 clinic in the United States.
Pre-assignment Details: This study consisted of two treatment periods. Following a Screening Period of 21 days, eligible participants were randomized in a 1:1 ratio to 1 of 2 treatment groups. Treatment Group A received efavirenz once daily on Day 1 and continued the regimen through Day 35 and a single dose of quizartinib on Day 15. Treatment Group B received a single dose of quizartinib on Day 1.
Period: Overall Study
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10.05) | 38.7 (10.22) | 39.6 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 15 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) Following Single Dose of Quizartinib With or Without Efavirenz
Description: Maximum Plasma Concentration (Cmax) is defined as the maximum observed plasma concentration and was an observed value for the study. Cmax was assessed for Quizartinib and active metabolite AC886.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 288, 360, 432, and 504 hours post-quizartinib dose
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set except for 1 participant from the Efavirenz 600 mg + Quizartinib 60 mg group due to insufficient data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Number analyzed (Participants) | 15 | 16
ng/mL
  Quizartinib | 130.0 (36.1) | 238.0 (76.9)
  AC886 | 11.0 (5.35) | 34.4 (18.2)
Statistical Analysis 1: Comparison: Efavirenz 600 mg + Quizartinib 60 mg vs Quizartinib 60 mg; Statistical comparison was analyzed for Quizartinib; Test type: Other — Least squares (LS) means were calculated from an analysis of variance (ANOVA) model on log-transformed scale. The LS means for each treatment were back transformed from the log scale to provide estimates of the geometric means (GMS). The ratio (%) of GMS was calculated and 90% Confidence Intervals (CIs) for the ratio (%) of GMS were presented; Ratio (%) of Geometric LS Mean = 55.24, 90% CI 2-sided [45.24 to 67.46] — For the comparison, the Efavirenz + Quizartinib treatment group represents the numerator and Quizartinib only treatment group represents the denominator
Statistical Analysis 2: Comparison: Efavirenz 600 mg + Quizartinib 60 mg vs Quizartinib 60 mg; Statistical comparison was analyzed for AC886; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 32.37, 90% CI 2-sided [23.79 to 44.05] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) Following Single Dose of Quizartinib With or Without Efavirenz
Description: Time of Maximum Plasma Concentration (Tmax) is defined as time of maximum observed plasma concentration and was an observed value from the study. Tmax was assessed for Quizartinib and active metabolite AC886.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 288, 360, 432, and 504 hours post-quizartinib dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Number analyzed (Participants) | 15 | 16
hours
  Quizartinib | 2.0 [2.0 to 4.0] | 4.0 [2.0 to 4.2]
  AC886 | 4.0 [2.0 to 4.0] | 4.0 [4.0 to 24.0]

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve up to the Last Quantifiable Concentration Post-Dose (AUClast) Following Single Dose of Quizartinib With or Without Efavirenz
Description: Area Under the Plasma Concentration-Time Curve up to the Last Quantifiable Concentration Post-Dose (AUClast) is defined as AUC from time 0 to the last measurable concentration, as calculated by the linear up-log down trapezoidal method and was calculated using non-compartmental analysis. AUClast was assessed for Quizartinib and active metabolite AC886.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 288, 360, 432, and 504 hours post-quizartinib dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Number analyzed (Participants) | 15 | 16
ng*h/mL
  Quizartinib | 2730 (1160) | 23600 (8420)
  AC886 | 185 (177) | 4110 (1320)
Statistical Analysis 1: Comparison: Efavirenz 600 mg + Quizartinib 60 mg vs Quizartinib 60 mg; Statistical comparison was analyzed for Quizartinib; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 11.11, 90% CI 2-sided [8.47 to 14.56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Efavirenz 600 mg + Quizartinib 60 mg vs Quizartinib 60 mg; Statistical comparison was analyzed for AC886; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 3.67, 90% CI 2-sided [2.47 to 5.45] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve up to Infinity (AUCinf) Following Single Dose of Quizartinib With or Without Efavirenz
Description: Area Under the Plasma Concentration-Time Curve up to Infinity (AUCinf) is defined as area under the plasma concentration-time curve from the time of dosing extrapolated to infinity and was calculated using non-compartmental analysis. AUCinf was assessed for Quizartinib and active metabolite AC886.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 288, 360, 432, and 504 hours post-quizartinib dose
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set except for 1 participant from the Efavirenz 600 mg + Quizartinib 60 mg group due to insufficient data. Data from participants where AUCinf based on extrapolation was greater than 20% was also excluded from the Efavirenz 600 mg + Quizartinib 60 mg group and Quizartinib 60 mg group.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Number analyzed (Participants) | 15 | 16
ng*h/mL
  Quizartinib: number analyzed (Participants) | 15 | 15
  Quizartinib | 2760 (1170) | 26000 (9880)
  AC886: number analyzed (Participants) | 14 | 15
  AC886 | 208 (183) | 4540 (1410)
Statistical Analysis 1: Comparison: Efavirenz 600 mg + Quizartinib 60 mg vs Quizartinib 60 mg; Statistical comparison was analyzed for Quizartinib; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 10.29, 90% CI 2-sided [7.73 to 13.70] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Efavirenz 600 mg + Quizartinib 60 mg vs Quizartinib 60 mg; Statistical comparison was analyzed for AC886; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 3.88, 90% CI 2-sided [2.62 to 5.76] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Terminal Half-Life (t1/2) Following Single Dose of Quizartinib With or Without Efavirenz
Description: Terminal Elimination Half-Life (t1/2) is defined as terminal elimination half-life and was calculated using non-compartmental analysis. AUClast was assessed for Quizartinib and active metabolite AC886. Half-life (t1/2) was assessed for Quizartinib and active metabolite AC886.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 288, 360, 432, and 504 hours post-quizartinib dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Number analyzed (Participants) | 15 | 16
hours
  Quizartinib | 23.8 (7.4) | 136 (40.1)
  AC886 | 11.9 (5.5) | 135 (33.5)

6. Primary Outcome: Metabolite to Parent Ratio (MPR) Based on Area Under the Curve for Active Metabolite AC886 Following Single Dose of Quizartinib With or Without Efavirenz
Description: AUCinf is defined as area under the plasma concentration-time curve from the time of dosing extrapolated to infinity and AUClast is defined as AUC from time 0 to the last measurable concentration, as calculated by the linear up-log down trapezoidal method. MPR is defined as a metabolite to parent ratio with metabolite as the numerator and the parent as the denominator. MPR corrected for molecular weight of AC886 of AUCinf and AUClast are reported and were calculated using non-compartmental analysis.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 288, 360, 432, and 504 hours post-quizartinib dose
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set except for 1 participant from the Efavirenz 600 mg + Quizartinib 60 mg group due to insufficient data. Data from participants where AUCinf based on extrapolation was greater than 20% was also excluded from MPR AUCinf.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Number analyzed (Participants) | 15 | 16
ratio
  MPR AUClast | 0.0675 (0.0403) | 0.186 (0.0753)
  MPR AUCinf: number analyzed (Participants) | 14 | 15
  MPR AUCinf | 0.0762 (0.0395) | 0.1880 (0.0777)

7. Primary Outcome: Total Apparent Clearance (CL/F) for Quizartinib Following Single Dose of Quizartinib With or Without Efavirenz
Description: Total Apparent Clearance (CL/F) is defined as total apparent clearance and was calculated using non-compartmental analysis.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 288, 360, 432, and 504 hours post-quizartinib dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Number analyzed (Participants) | 15 | 16
L/h | 12.210 (7.6937) | 1.1849 (0.51388)

8. Primary Outcome: Volume of Distribution in the Terminal Phase (Vz/F) for Quizartinib Following Single Dose of Quizartinib With or Without Efavirenz
Description: Volume of Distribution in the Terminal Phase (Vz/F) is defined as volume of distribution in the terminal phase and was calculated using non-compartmental analysis.
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 288, 360, 432, and 504 hours post-quizartinib dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Number analyzed (Participants) | 15 | 16
L | 359.9 (102.23) | 214.9 (59.82)

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Following Single Dose of Quizartinib With or Without Efavirenz
Description: A Treatment-Emergent Adverse Events (TEAE) is defined as any event not present prior to the initiation of the drug treatment of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment. Number of any TEAE that is related and unrelated to study medication is presented.
Time Frame: Baseline up to 30 days post last dose, up to approximately 2 months
Population: TEAEs were assessed using the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
Number analyzed (Participants) | 16 | 16
Participants | 13 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of signing the informed consent form up to 30 days after last dose, up to 2 months.
Description: Adverse events were defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All-cause mortality includes all deaths that occurred during the study and within the 30 days after the last dose of the study drug.
Arm/Group | Efavirenz 600 mg + Quizartinib 60 mg | Quizartinib 60 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 13/16 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efavirenz 600 mg + Quizartinib 60 mg (N=16) | Quizartinib 60 mg (N=16)
Headache (Nervous system disorders) | 6 | 2
Dizziness (Nervous system disorders) | 5 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Vessel puncture site pain (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Eyelid irritation (Eye disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Syphilis (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT04459598/Prot_SAP_000.pdf